CLINICAL TRIAL: NCT03911843
Title: Omega 3 Long Chain Polyunsaturated Fatty Acids, Enriched Mediterranean Diet and Vitamin D Supplementation in Childhood Type 1 Diabetes: One Year Case-cohort Study
Brief Title: Omega-3 and Vitamin D Supplements in Childhood T1D
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Collaborators: University of Eastern Piedmont (Other)
Responsible Party: Principal Investigator, Francesco Cadario, MD, MD Division of Pediatrics, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AOU Novara
Record Dates: First submitted 2019-03-18; First posted 2019-04-11 (Actual); Results first posted 2021-03-23 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: omega3; T1D remission period; honeymoon period; AA/EPA ratio
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: A cohort study was performed in 2017, in all T1D patients 1-18 years old with onset in the years 2014-2017. Supplementation with omega3 was proposed to all subjects with onset in 2017. Patients with onset in 2014-2015-2016 were enrolled only as control subjects. The work was performed on retrospectively collected data in medical records for patients with start of the disease in 2014-2016. Patients enrolled since 2017 have been studied prospectively.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CASES (Experimental): Of eligible subjects, 26/64 started an intervention program with Ω-3 (CASES). The intervention consisted in supplementation with highly purified Ω-3, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) at a dose of 50-60 mg/kg/day for 12 months
  Interventions: Drug: omega-3 supplementation; Drug: Vitamin D supplementation
- CONTROLS (Active Comparator): Others 38/64 subjects joined to the study as data contributors, and were entered as controls (CONTR).
  Interventions: Drug: Vitamin D supplementation

INTERVENTIONS:
Drug: omega-3 supplementation — Supplementation with Ω-3, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) at a dose of 50-60 mg/kg/day for 12 months, currently underway or completed after 12 months of omega-3 administration, in 22/64 T1D children
  Other Names: Ener Zone Omega 3 RX® Equipe Enervit
  Arms: CASES
Drug: Vitamin D supplementation — Cholecalciferol 1000 IU/die

SUMMARY:
The study was conducted in 64 patients with T1D of which 26 had the onset in 2017, and 38 in 2016, 2015 and 2014. All received vitamin D 1000 IU /day since disease's onset. Moreover in the 2017 group omega-3 were supplemented, starting within 3 and 6 months from the disease's outbreak, and those were considered cases; the other 38 were enrolled as controls. Four cases and one control dropped out. Finally in 59/64 were compared data of glycosylated hemoglobin percentage (HbA1c%), average insulin daily requirement (IU/Kg/day), and IDAA1c [Insulin Daily dose Adjusted for HbA1c, a surrogate index of residual endogen insulin secretion, calculated as insulin daily dose (IU/Kg/24 h) x 4 + HbA1c%] at recruitment (T0), and 3 (T3), 6 (T6), 12 (T12) months after. T0 in cases was at the start of supplementation of omega-3, and consequently 3, 6 and 12 months after; in controls were found data in clinical records of outpatient beginning from the 3rd month and 3-6-12 months thereafter. Then 22 cases and 37 controls were compared.

DETAILED DESCRIPTION:
Was assessed the comparability of cases and controls at baseline for gender, age, body weight, HbA1c% and device for insulin therapy.

The preparation of omega-3 administered was a highly purified fish oil to avoid pollutants, containing a mixture of omega-3 long chain fatty acids standardized for contents of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) in a 2: 1 ratio, in capsules or in liquid form. The liquid preparation was used in the case of difficulties in swallowing capsules or concomitant celiac disease because it was certified as gluten-free (Ener Zone Omega 3 RX® Equipe Enervit). The preparations contained antioxidants to preserve omega-3 LCFA, tocopherol (1 mg in 1 g of omega-3 LCFA), palmitate, and rosemary extract. EPA and DHA were administered at 50-60 mg/kg/day for 12 months. The investigation of Arachidonic Acid (AA)/EPA ratios was performed in cases on recruitment (T0), and repeated after 3 (T3), 6 (T6), and 12 months (T12).

Cholecalciferol supplementation was fixed at 1000 IU/day (25 mcg/day), both in cases and controls. Vitamin D level was determined as 25(OH)D level at the clinical onset of T1D, at T0, T3, T6, and T12 in cases, and at clinical onset of controls.

ELIGIBILITY:
Inclusion Criteria:

* All T1D patients aged 1-18 years whose disease onset had been in 2017, 2016, 2015, 2014 affering to the Pediatric Diabetology of AOU Novara (Italy)
* written consents of parents
* without assumption of omega 3 supplementation before 2017

Exclusion Criteria:

* renal cysts
* sarcoidosis
* histoplasmosis
* hyperparathyroidis
* lymphoma
* tuberculosis
* Patients treated with drugs that could affect immunity or glucose metabolism, including corticosteroids, ciclosporin and tacrolimus

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cadario, MD, Principal Investigator — Pediatric Clinic of AOU Novara

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in the publication will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: the IPD and any additional supporting information will become available and for ten years, including the start and end dates or period of availability. This may be provided starting to date when data are published or otherwise made available.
Access Criteria: adress the request to Central Contact Person

REFERENCES:
- [Background] Cadario F, Savastio S, Ricotti R, Rizzo AM, Carrera D, Maiuri L, Ricordi C. Administration of vitamin D and high dose of omega 3 to sustain remission of type 1 diabetes. Eur Rev Med Pharmacol Sci. 2018 Jan;22(2):512-515. doi: 10.26355/eurrev_201801_14203. PMID 29424911
- [Background] Baidal DA, Ricordi C, Garcia-Contreras M, Sonnino A, Fabbri A. Combination high-dose omega-3 fatty acids and high-dose cholecalciferol in new onset type 1 diabetes: a potential role in preservation of beta-cell mass. Eur Rev Med Pharmacol Sci. 2016 Jul;20(15):3313-8. PMID 27467009
- See also: Pilot Study of OMEGA-3 and Vitamin D in High-Dose in Type I Diabetic Patients (POSEIDON) — http://clinicaltrials.gov/ct2/show/NCT03406897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started 03/17/2017 with the enrollment of the first patient, and ended on 06/08/2019 with the end of the omega-3 supplementation period of the last enrolled patient. All participants were introduced since the beginning of T1D to tailored insulin therapy, to Mediterranean diet (according to a standardized item detailed in reference), and received 1000 IU/day of vitamin D supplementation.
Groups:
- CASES New T1D Onsets 2017: All the New T1D Onsets 2017 received a further supplementation of ultra refined fish oil, enriched in LC-PUFA omega 3, containing standardized concentrations EPA + DHA (2:1), at 60 mg/kg/day. The supplementation with omega 3 started within 3th and 6th months after the clinical T1D onset and lasted one year.
- CONTROLS Previous T1D Onsets: All Previous T1D Onsets (2014-2016) receiving vitamin D and Mediterranean diet without omega 3 supplementation, were continuously recruited. Retrospectively their available data from 3th and 6th months from the clinical onset to T1D, for the following year, were compared.
Period: Overall Study
Arm/Group | CASES New T1D Onsets 2017 | CONTROLS Previous T1D Onsets
Started | 26 | 38
Completed | 22 | 37
Not Completed | 4 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only the subjects who finished the study contributed to the result
Groups:
- CASES: The T1D onsets were eligible subjects, of which 26/64 new onsets started an intervention program with Ω-3 (CASES). The intervention consisted in supplementation with highly purified Ω-3, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) at a dose of 60 mg/kg/day for 12 months. The supplementation with omega 3 started within 3th and 6th months of T1D clinical onset and lasted one year.
  They had been introduced to the Mediterranean diet according to a standardized item and received 1000 IU/day of vitamin D supplementation since the beginning of T1D
- CONTROLS: The Previous T1D onsets, 38/64 subjects joined to the study as controls (CONTROLS). They received vitamin D supplementation 1000 IU/day and Mediterranean diet according to a standardized item since the onset of T1D, without omega 3; retrospectively their available data from 3th and 6th months of overt disease for the following year, were compared
- Total: Total of all reporting groups
Arm/Group | CASES | CONTROLS | Total
Number analyzed (Participants) | 26 | 38 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 38 | 64
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (4.6) | 8.8 (3.6) | 8.75 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 12 | 18 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Italian | 20 | 33 | 53
  North Africa | 4 | 4 | 8
  Albania | 1 | 1 | 2
  Pakistan | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Italy | 26 | 38 | 64

OUTCOME MEASURES:

1. Primary Outcome: Daily Insulin Need (IU/Kg/Day) and Daily Insulin Pre-meal Demand (Pre-meal IU/Kg/Day) at 12 Months
Description: The Daily Insulin Needs (IU/Kg/day), and the Daily Insulin Pre-meal Demand (Pre-meal IU/Kg/day) respectively represent the average total (sum of boluses and basal) and average pre-meal (sum of pre-meal boluses) insulin doses administered in one day to each patient.
  They have been calculated over a week, and were expressed in International Units / Kg of weight, higher values mean a worse outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: IU/Kg/day
Arm/Group | CASES New T1D Onsets 2017 | CONTROLS Previous T1D Onsets
Number analyzed (Participants) | 22 | 37
IU/Kg/day
  Daily insulin need | 0.49 (0.2) | 0.63 (0.1)
  Daily Insulin Pre-meal Demand | 0.22 (0.1) | 0.34 (0.1)
Statistical Analysis 1: Comparison: CASES New T1D Onsets 2017 vs CONTROLS Previous T1D Onsets; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — the p-value of significance was calculated using the analysis system; Mean Difference (Net) = -0.14
Statistical Analysis 2: Comparison: CASES New T1D Onsets 2017 vs CONTROLS Previous T1D Onsets; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.14

2. Primary Outcome: HbA1c Percentage
Description: percentage of glycated hemoglobin measured through the high-performance liquid chromatography (HPLC).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | CASES New T1D Onsets 2017 | CONTROLS Previous T1D Onsets
Number analyzed (Participants) | 22 | 37
percentage of HbA1c | 7.4 (1) | 7.8 (1)
Statistical Analysis 1: Comparison: CASES New T1D Onsets 2017 vs CONTROLS Previous T1D Onsets; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Number of Participants With Insulin Demand Adjusted for HbA1c %(IDAA1c) <9
Description: The IDAA1c (insulin daily dose adjusted for glycosylated hemoglobin percentage) was calculated as HbA1c percentage + average daily insulin dose (IU/kg/24 h) x 4. A score <9 meet definition of partial remission and Residual Endogenic Insulin Secretion (REIS). IDAA1c represents a surrogate index of insulin secretion and of metabolic control. In a scale from 5 to 12, higher score mean a worse outcome (e.g. <5.5 is expected in a normal individual, <9 in an individual in partial remission. See reference).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | CASES New T1D Onsets 2017 | CONTROLS Previous T1D Onsets
Number analyzed (Participants) | 22 | 37
Participants | 12 | 7
Statistical Analysis 1: Comparison: CASES New T1D Onsets 2017 vs CONTROLS Previous T1D Onsets; Test type: Superiority; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: The observation interval of side effects was in each case into the period of omega-3 supplementation (T0-T12), lasting 12 months, and into a comparable period in the controls.
Description: 1. Chronic diarrhea lasting 2 weeks of duration in a female case. The administration of supplementation with omega 3 was interrupted
  2. Isolated thyrotropine deficiency, in a teenager girl with pre-existing autoimmune thyroiditis. The administration of supplementation with omega 3 was interrupted
  3. Activated partial thromboplastin time (observable entity) without clinical symptoms observed. At the end of the study, one year after the start of omega 3 supplementation
Groups:
- CASES New T1D Onsets 2017: All the New T1D Onsets 2017 received Mediterranean diet, vitamin D 1000 IU/day, and a further supplementation of ultra refined fish oil, enriched in LC-PUFA omega 3, containing standardized concentrations EPA + DHA (2:1), at 60 mg/kg/day. The supplementation with omega 3 started within 3th and 6th months after the clinical T1D onset and lasted one year.
Arm/Group | CASES New T1D Onsets 2017 | CONTROLS Previous T1D Onsets
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/37
Other Adverse Events (participants affected / at risk) | 1/26 | 0/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CASES New T1D Onsets 2017 (N=26) | CONTROLS Previous T1D Onsets (N=38)
persistent diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — the diarrhea started soon after the start of omega 3 supplementation, that was interrupted. The diarrhea lasted 2 weeks
transient suppression of TRH (Endocrine disorders) | 1 (1) | 0 (0) — in one teenager girl with pre-existing autoimmune thyroiditis, a transient suppression of TRH was found, lasting 3 months after omega 3 suspension
an extension of the aPTT clotting (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — an extension of the aPTT clotting time at the end of the supplementation period was verified.

LIMITATIONS AND CAVEATS:
The study was not randomized and Controls were retrospective, whereby the comparability between Cases and Controls concerned only HbA1c percentage, Daily Insulin Needs (IU/Kg/day) and IDAA1c, indirect indices of residual endogen insulin secretion (REIS)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT03911843/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT03911843/SAP_001.pdf
  • Informed Consent Form (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT03911843/ICF_002.pdf